CLINICAL TRIAL: NCT01534559
Title: A Pharmacist-led Medicines Management Outpatient Service for Patients at High Risk of Medication Related Problems
Brief Title: Pharmacist-led Medicines Management Outpatient Service
Acronym: MMC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, James McElnay, Chief Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUB B11/34
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Patients at High Risk of Medicine-related Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Outpatient Medicine Management Clinic (Experimental): Consented patients will attend two outpatient clinic appointments to receive help with any (potential) medicine-related problems
  Interventions: Other: Medicines Management Outpatient service
- Control (No Intervention): Patients will receive the normal care provided by the hospital

INTERVENTIONS:
Other: Medicines Management Outpatient service — New customised clinical pharmacy service (medicines management clinic and follow-up phone calls)
  Other Names: Medicines Management Clinic; Pharmacist-led outpatient service
  Arms: Outpatient Medicine Management Clinic

SUMMARY:
It widely accepted that a number of medication related problems can occur after the patient has been discharged from the hospital. An obvious extension of the ongoing integrated medicines management programme (IMMP) is therefore to provide a medicines management clinic within an outpatient setting as well as follow-up telephone calls from a clinical pharmacist. This study aims to assess the influence a pharmacist-led medicines management outpatient service on patients at high risk of medication related problems.

It is anticipated that this service will

* Ensure continuity of pharmaceutical care for patients post discharge.
* Reinforce patient education in order to improve knowledge and understanding of the medication prescribed.
* Ensure that both prescription medicines and OTC preparations are used appropriately.
* Facilitate the communication with other members of healthcare team in order to agree and implement measures to overcome medication related problems.

DETAILED DESCRIPTION:
Patient safety and wellbeing are central concerns within the health service. Recent publications have highlighted the importance of medicines management and have called for local strategies to be introduced. An Integrated Medicines Management Programme (IMMP) has been implemented within Northern Health and Social Care Trust to ensure that a co-ordinated pharmacy service is available throughout the hospital stay for its medical patients. The IMMP has resulted in a number of benefits including improved patient safety, more effective use of medications, reduced length of stay, reduced readmissions rates, improved communication across the healthcare interface and user satisfaction.

It is widely accepted that a number of medication related problems can occur post discharge when complicated medication regimens can often prove confusing. This can lead to mismanagement of medicines and early rehospitalisation of patients. Although these problems are frequently commented upon, research in this area is still lacking. The present project aims to examine an extension of the present IMM service by evaluating the impact/patient benefit of a customised outpatient service provided by clinical pharmacy staff to patients post-discharge. An increase in patients' medicines adherence, a greater satisfaction with information about their medicines, improved beliefs about the necessity of their medicines, a decrease in medicines-related problems, a decrease in re-hospitalisation rates, extended time to re-hospitalisation, and a decrease in overall costs of patients care is anticipated.

This study will be carried out as a collaboration between the School of Pharmacy at Queen's University Belfast and the Northern Health and Social Care Trust (2 sites; Antrim Area Hospital and Whiteabbey Hospital).

ELIGIBILITY:
Inclusion Criteria:

Patients (>= 18 years old) admitted into one of the study hospitals as acute/unscheduled medical admission and meet at least one of the following criteria:

* Prescribed five or more regular long term medications.
* Have three or more changes to medications during hospital stay.
* Past history of medication related problems.
* Patient referred to the medicines management clinic service by hospital doctor or clinical pharmacist due to concerns about ability to manage medicines in primary care.

Exclusion Criteria:

* Patient being discharged to residential/nursing homes
* Palliative care patients
* Patients unable to give informed consent e.g. Alzheimer's Disease
* Patients unable to use telephone at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Time to readmission to hospital | Over 12 month post discharge

SECONDARY OUTCOMES:
Number of Readmission | Over 12 months post discharge
Number of GP consultations and GP home visits | over 12 month post discharge
Number of Accident and Emergency (A&E) visits | over 12 month post discharge
Medication Appropriateness Index (MAI) score | Will be assessed at dischrge and 4, 8 and 12 month post discharge
Health-related quality of life (HRQOL) | Over 12 months post discharge, every 4 months
  This will be assessed using EQ-5D questionnaire
Medication Adherence Assessments; | Over 12 month post discharge. Every 4 months.
  Adherence will be assessed using the medication adherence report scale (MARS). Beliefs about medicines will be assessed using the validated beliefs about medicines questionnaire (BMQ).
Cost Utility Analysis | Over 12 month post discharge.

CONTACTS AND LOCATIONS:
Overall Officials: James C McElnay, BSc, PhD, Study Chair — Queen's University, Belfast; Michael G Scott, BSc, PhD, Principal Investigator — Northern Health and Social Care Trust
Locations (1):
- Northern Health and Social Care Trust, Antrim, Northern Ireland, United Kingdom